CLINICAL TRIAL: NCT01662518
Title: A Safety and Efficacy Study to Assess DDS-25 Gauge in Patients With Macular Edema Secondary to Retinal Vein Occlusion (RVO)
Brief Title: DDS-25 Gauge in Patients With Macular Edema Secondary to Retinal Vein Occlusion (RVO)
Acronym: DDS-25
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centro de Pesquisa Rubens Siqueira (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rubens Camargo Siqueira, MD,PhD - Principal Investigator, Centro de Pesquisa Rubens Siqueira
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bramets-01
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion

STUDY DESIGN:
Intervention Model Description: intervention group: 25-gauge biodegradable implant containing 350 μg of dexamethasone (DDS-25) for the treatment of decreased vision due to macular edema associated with central or branch retinal vein occlusion.
Oversight: Data Monitoring Committee: No

ARMS (1):
- DDS-25 (Experimental): Intravitreal injection of DDS-25(Dexamethasone drug delivery system )
  Interventions: Device: Dexamethasone drug delivery system (DDS-25)

INTERVENTIONS:
Device: Dexamethasone drug delivery system (DDS-25) — 350 mg Dexamethasone posterior segment drug delivery system (DDS-25) injection into the vitreous cavity at baseline

SUMMARY:
This study will evaluate the safety and efficacy of an intravitreal implant of dexamethasone (DDS-25) for the treatment of macular edema associated with retinal vein occlusion.

DETAILED DESCRIPTION:
Evaluate the effects on visual acuity, electroretinography, fluorescein angiography and optical coherence tomography in 10 patients with macular edema associated with retinal vein occlusion undergoing intravitreal injection of implant of dexamethasone (DDS-25).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with macular edema resulting from retinal vein occlusion
* Decrease in visual acuity in at least one eye as a result of macular edema (20/50 or worse)
* Visual acuity in other eye no worse than 20/200

Exclusion Criteria:

* Known anticipated need for ocular surgery within next 12 months
* History of glaucoma or current high eye pressure requiring more than 1 medication
* Diabetic retinopathy
* Uncontrolled systemic disease
* Known steroid-responder
* Use of systemic steroids
* Use of warfarin/heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-07; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | Day 0 - Day 180

SECONDARY OUTCOMES:
Change in central foveal thickness at 48 weeks | 1 day to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rubens C Siqueira, MD,PhD, Principal Investigator — Centro de Pesquisa Rubens Siqueira
Locations (1):
- Centro de Pesquisa Rubens Siqueira, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Retin Cases Brief Rep. 2016 Sep 14. [Epub ahead of print] SAFETY AND FEASIBILITY OF A NOVEL 25-GAUGE BIODEGRADABLE IMPLANT OF DEXAMETHASONE FOR TREATMENT OF MACULAR EDEMA ASSOCIATED WITH RETINAL VEIN OCCLUSION: A PHASE I CLINICAL TRIAL.
  Cunha RB1, Siqueira RC, Messias A, Scott IU, Fialho SL, Cunha-Junior AD, Jorge R.

REFERENCES:
- See also: SAFETY AND FEASIBILITY OF A NOVEL 25-GAUGE BIODEGRADABLE IMPLANT OF DEXAMETHASONE FOR TREATMENT OF MACULAR EDEMA ASSOCIATED WITH RETINAL VEIN OCCLUSION: A PHASE I CLINICAL TRIAL. — http://www.ncbi.nlm.nih.gov/pubmed/27632583